CLINICAL TRIAL: NCT05113667
Title: Impact of Clinical Pharmacist-led Appropriate Acid Suppression Therapy Stewardship Program on Hospitalized Older Patients: A Non-Randomized Controlled Study
Brief Title: Clinical Pharmacist-led Appropriate Acid Suppression Therapy Stewardship Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Betul Okuyan, Assoc.Prof., Marmara University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MUHSI-2019/29-78
Record Dates: First submitted 2021-10-17; First posted 2021-11-09 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Geriatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical pharmacist-led services (Experimental): Clinical Pharmacist-led Appropriate Acid Suppression Therapy Stewardship Program
  Interventions: Other: Clinical Pharmacist-led Appropriate Acid Suppression Therapy Stewardship Program
- Control group (No Intervention): Usual care

INTERVENTIONS:
Other: Clinical Pharmacist-led Appropriate Acid Suppression Therapy Stewardship Program — Clinical pharmacist provided medication reconciliation and medication review during the hospital stay.
  Arms: Clinical pharmacist-led services

SUMMARY:
To evaluate the impact of clinical pharmacist-led appropriate acid suppression therapy stewardship program in hospitalized older patients.

DETAILED DESCRIPTION:
This prospective, nonrandomized controlled study was conducted in older patients who ordered proton pump inhibitor (PPI) at admission in an internal medicine service of tertiary training and research hospital. In the intervention group, clinical pharmacist-led services (including medication reconciliation and medication review) were conducted during hospitalization and at discharge by using the guidelines and potentially inappropriate medications (PIM) criteria [American Geriatric Society-AGS Beers Criteria©, 2019]. Medication Appropriateness Index (MAI), inappropriate PPI cost, and hospitalization for gastrointestinal bleeding within 1 year after discharge were calculated in both groups

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or greater
* Admitted to the hospital with any reason
* Ordered at least one PPI dose within 48 hours of admission

Exclusion Criteria:

* Transferred to another ward (including an intensive care unit)
* Having active gastrointestinal bleeding
* Having active malignity

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Appropriateness of Proton Pump Inhibitors Usage | during hospital stay, an average of 14 days
  The rate of appropriateness use of proton pump inhibitors based on the guidelines at hospital stay
Potentially Inappropriate Proton Pump Inhibitors Usage | at discharge, an average of 14 days after admission to hospital
  The rate of potentially inappropriate use of proton pump inhibitors based on American Geriatric Society Beers Criteria© 2019

SECONDARY OUTCOMES:
Clinical outcome | 1 year
  The number of patients who hospitalized for bleeding within 1 year after discharge
Cost saving during hospital stay | during hospital stay, an average of 14 days
  Medication cost for inappropriate PPI during hospital study
Medication Appropriateness Index for Proton Pump Inhibitors at hospital stay | during hospital stay, an average of 14 days
  Medication Appropriateness Index (MAI); included 10 items. Each item was weighted from 1-3. The highest score per medication was 18.
  Higher scores of this index represent more inappropriateness of each medication.
Cost saving after discharge | a month
  Medication cost for potentially inappropriate PPI after discharge
Medication Appropriateness Index for Proton Pump Inhibitors at discharge | at discharge, an average of 14 days after admission to hospital
  Medication Appropriateness Index (MAI); included 10 items. Each item was weighted from 1-3. The highest score per medication was 18.
  Higher scores of this index represent more inappropriateness of each medication.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Okuyan, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dumlu HI, Sancar M, Ozdemir A, Okuyan B. Impact of a clinical pharmacist-led stewardship program for the appropriate use of acid suppression therapy in older hospitalized patients: a non-randomized controlled study. Int J Clin Pharm. 2022 Aug;44(4):914-921. doi: 10.1007/s11096-022-01394-8. Epub 2022 Apr 21. PMID 35449351